CLINICAL TRIAL: NCT04113447
Title: Mitochondrial Donation: An 18 Month Outcome Study.
Status: Recruiting | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 8075
Record Dates: First submitted 2018-08-13; First posted 2019-10-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: observational — observational

SUMMARY:
The Investigator proposes to record the fetal and postnatal development of children conceived using Mitochondrial Donation (MD) and to perform expert assessment of development at 18 months (corrected for gestational age) using the internationally validated Bayley-III developmental assessment tool.

DETAILED DESCRIPTION:
To record the fetal and postnatal development of children conceived using Mitochondrial Donation and to perform internationally validated Bayley-III developmental assessment tool at 18 months (corrected for gestational age).

The null hypothesis for this research is that children born following the use of Mitochondrial Donation (IVF) techniques have normal neurodevelopment developmental outcomes at 18 months.

ELIGIBILITY:
Inclusion Criteria:

Women will only be eligible if they meet all of the following criteria.

* Women with confirmed mtDNA mutation
* Suitable to undergo Mitochondrial Donation as a treatment (in line with HFEA license)
* Informed Consent for the study obtained before Mitochondrial Donation treatment commences
* Ability and willingness to adhere to the protocol including evaluation schedule
* Willingness to make available information collected during pregnancy, delivery and up to the child's age of 18 months (corrected for gestational age)

Exclusion Criteria:

Women will not be eligible if they meet any of the following criteria

* Declined Mitochondrial Donation as a treatment (in line with HFEA license)
* Inability or unwillingness to adhere to the protocol including evaluation schedule
* Unwillingness to make available information collected during pregnancy, delivery and up to the child's age of 18 months (corrected for gestational age)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with mitochondrial disease undergoing mitochondrial donation treatment
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
A normal neurodevelopmental quotient scored using a Bayley-III ( Bayley Scales of Infant and Toddler Development, Third Edition) at 18 months (corrected | 18 months
  The Bayley Scale of Infant and Toddler Development, Third Edition (Bayley III) measures physical, motor, sensory, and cognitive development in babies and young children. The scale encompasses five developmental domains - cognitive, language, motor, social-emotional and adaptive behaviour. The structure of the Bayley-III Scales allows clinicians to administer each of the five scales (cognitive, language-receptive and expressive, motor-fine and gross, social-emotional, and adaptive behaviour) independent of others. Higher scores in each scale indicates more advanced development. Performance is summarised via scaled scores for each subtest, and composite scores for each scale, together with percentile ranks, developmental age equivalents, and growth scores. Discrepancy information is used to determine whether there are significant differences between a child's abilities in the domains measured, and how prevalent these differences are in the norming sample. A total score is not provided.

SECONDARY OUTCOMES:
1)Normal hearing as assessed by formal audiology, | 18 months
  Formal Audiology
2)Normal vision as assessed by ophthalmologist | 18 months
  Ophthalmology Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No